CLINICAL TRIAL: NCT05493735
Title: Lidocaine for Pessary Removal and Reinsertion Pain Reduction
Brief Title: Lidocaine for Pessary Check Pain Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro004522
Record Dates: First submitted 2022-07-15; First posted 2022-08-09 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence
Keywords: Pessary; Lidocaine; Pain Reduction; Pessary Check; Pessary Removal; Pessary Reinsertion; Lubricating Jelly
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress | interventions — Lidocaine; Gels

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Lubricating jelly (placebo) will be placed in the vagina to the level of the pessary, five minutes prior to pessary removal.
  Interventions: Drug: Placebo Jelly
- Experimental (Experimental): Lidocaine jelly will be placed in the vagina to the level of the pessary, five minutes prior to the pessary removal.
  Interventions: Drug: Lidocaine Hcl 2% Jelly

INTERVENTIONS:
Drug: Lidocaine Hcl 2% Jelly — Participants in the experimental arm will undergo pessary removal and reinsertion after the application of lidocaine topical gel.
  Other Names: Lidocaine Jelly
  Arms: Experimental
Drug: Placebo Jelly — Participants in the control arm will undergo pessary removal and reinsertion after the application of lubricating jelly.
  Other Names: Lubricating Gel; Vaginal Lubricant
  Arms: Control

SUMMARY:
The primary objective of this study is to estimate the effect of lidocaine jelly on patient pain at the time of office pessary removal.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of lidocaine jelly on patient pain at the time of office pessary removal and reinsertion. All patients presenting to the University of South Florida Urogynecology clinic for a pessary maintenance appointment or "pessary check" will be screened as potential study participants. After being informed of risks and benefits of participation, informed consent will be obtained. Patients will be randomized into two groups: the control group or experimental group. The patient will complete a brief questionnaire and pain assessment using a Visual Analog Scale (VAS).

Patients will be blinded. The investigators will be unblinded. The investigators will apply the jelly (lidocaine vs lubricating). The participant will have an equal chance of being in the control arm or experimental arm. After 5 minutes, the investigator will assess the patient's genital hiatus with valsalva and proceed with pessary removal per the investigator's routine. The patient will complete another VAS to indicate pain level after pessary removal. The investigator will perform a speculum exam per routine and then reinsert the pessary. The patient will complete a final VAS to indicate level of pain after pessary reinsertion along with a brief final questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Presenting for routine pessary management for prolapse, stress urinary incontinence, or both with a pessary in place
* able to provide written informed consent
* able to complete the visual analog scale

Exclusion Criteria:

* Women less than 18 years of age.
* Patients who speak neither English nor Spanish
* Pregnancy
* Medical contraindication to lidocaine
* Planned change in pessary size or type
* Patients who remove and reinsert their pessary at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in patient's pain using the visual analog scale (VAS) after pessary removal | 0 and 5 minutes
  Self-reported pain level at time of pessary removal controlling for baseline pain. Scale is from 0 to 10 (0=no pain and 10=worst pain)

SECONDARY OUTCOMES:
Change in patient's pain using the visual analog scale (VAS) after pessary reinsertion | 0 and 10 minutes
  Self-reported pain level at time of pessary reinsertion controlling for baseline pain. Scale is from 0 to 10 (0=no pain and 10=worst pain)
Genital Hiatus with Valsalva | 0 minutes
  Genital hiatus measurement in centimeters prior to removal of the pessary

CONTACTS AND LOCATIONS:
Overall Officials: Araba A Jackson, MD, Principal Investigator — University of South Florida
Locations (1):
- USF Health Outpatient Urogynecology Clinics, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donnelly MJ, Powell-Morgan S, Olsen AL, Nygaard IE. Vaginal pessaries for the management of stress and mixed urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Sep-Oct;15(5):302-7. doi: 10.1007/s00192-004-1163-7. Epub 2004 Aug 5. PMID 15300365
- [Background] Nguyen JN, Jones CR. Pessary treatment of pelvic relaxation: factors affecting successful fitting and continued use. J Wound Ostomy Continence Nurs. 2005 Jul-Aug;32(4):255-61; quiz 262-3. doi: 10.1097/00152192-200507000-00010. PMID 16030465
- [Background] Lone F, Thakar R, Sultan AH, Karamalis G. A 5-year prospective study of vaginal pessary use for pelvic organ prolapse. Int J Gynaecol Obstet. 2011 Jul;114(1):56-9. doi: 10.1016/j.ijgo.2011.02.006. Epub 2011 May 14. PMID 21575953
- [Background] Taege SK, Adams W, Mueller ER, Brubaker L, Fitzgerald CM, Brincat C. Anesthetic Cream Use During Office Pessary Removal and Replacement: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):190-197. doi: 10.1097/AOG.0000000000002098. PMID 28594757
- [Background] Keskin AE, Onaran Y, Duvan IC, Simavli S, Kafali H. Topical anesthetic (lidocaine-prilocaine) cream application before speculum examination in postmenopausal women. J Minim Invasive Gynecol. 2012 May-Jun;19(3):350-5. doi: 10.1016/j.jmig.2012.01.005. Epub 2012 Mar 13. PMID 22417905
- [Background] Ozel BZ, Sun V, Pahwa A, Nelken R, Dancz CE. Randomized controlled trial of 2% lidocaine gel versus water-based lubricant for multi-channel urodynamics. Int Urogynecol J. 2018 Sep;29(9):1297-1302. doi: 10.1007/s00192-018-3576-8. Epub 2018 Feb 17. PMID 29455237